CLINICAL TRIAL: NCT01745588
Title: Autologous Stem Cell Transplant With Pomalidomide (CC-4047®) Maintenance Versus Continuous Clarithromycin/ Pomalidomide / Dexamethasone Salvage Therapy in Relapsed or Refractory Multiple Myeloma: A Phase 2 Open-Label Randomized Study by Tristate Consortium
Brief Title: Autologous Stem Cell Transplant With Pomalidomide (CC-4047®) Maintenance Versus Continuous Clarithromycin/ Pomalidomide / Dexamethasone Salvage Therapy in Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Celgene Corporation (Industry); Weill Medical College of Cornell University (Other); North Shore University Hospital (Other); Rutgers Cancer Institute of New Jersey (Other); State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-138
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
Keywords: CC-4047(Pomalidomide)Pomalyst; Clarithromycin; Biaxin; DEXAMETHASONE; (ClaPD); Stem cell; 12-138
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Dexamethasone; Clarithromycin

ARMS (2):
- Clarithromycin + Pomalidomide + Dexamethasone + stem cell (Experimental): All patients will receive 4 cycles of clarithromycin 500mg twice daily on days 1-28, pomalidomide 4 mg daily on days 1 through 21 and dexamethasone orally at a dose of 40 mg daily on days 1, 8, 15, and 22 of each 28-day cycle. Patients randomized to auto-SCT will proceed within 28 days after completion of the 4th cycle of ClaPD to receive melphalan 140mg/m2 or 200mg/m2 (as per institutional guidelines) followed by hematopoietic cell infusion.
  Interventions: Drug: Pomalidomide; Procedure: stem cell; Drug: Clarithromycin
- Clarithromycin + Pomalidomide + Dexamethasone Alone (Experimental): All patients will receive 4 cycles of clarithromycin 500mg twice daily on days 1-28 pomalidomide 4 mg daily on days 1 through 21 and dexamethasone orally at a dose of 40 mg daily on days 1, 8, 15, and 22 of each 28 day cycle. Patients assigned to ClaPD alone will receive 5 additional cycles of ClaPD.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Clarithromycin

INTERVENTIONS:
Drug: Pomalidomide
Procedure: stem cell
  Arms: Clarithromycin + Pomalidomide + Dexamethasone + stem cell
Drug: Dexamethasone
  Arms: Clarithromycin + Pomalidomide + Dexamethasone Alone
Drug: Clarithromycin

SUMMARY:
The purpose of this study is to see whether pomalidomide (also known as Pomalyst) reduces the number of myeloma cells in the bones, and to see what is the best way to use pomalidomide in patients with myeloma. To do this, the investigators want to compare two types of treatment using pomalidomde. This is a randomized trial which means that the decision as to which treatment the patient will receive will be made by a computer, much like flipping a coin.

All patients start by receiving 4 cycles of clarithromycin, pomalidomide and dexamethasone (ClaPD). After 4 cycles, half of the patients will undergo an autologous stem cell transplant followed by pomalidomide (Group 1). The other half of the patients will continue to receive ClaPD for 9 cycles to be followed by pomalidomide maintenance. (Group 2).

At the end of the study, the two groups will be compared to see if there is a difference in disease outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed relapsed multiple myeloma as defined by the International Myeloma Working Group (IMWG).
* Patients must have measurable disease as defined by the International Uniform Response Criteria, defined as any of the following:
* serum M-protein of ≥ 500mg/dL
* urine M-protein of ≥ 200mg/ 24 hours
* involved free light chain ≥ 10mg/dL provided serum free light chain ratio is abnormal
* Patients must have had a previous auto-SCT performed as part of a consolidation of an initial remission and had a remission, defined as a partial response or greater that lasted at least 12 months either on or off maintenance therapy without evidence of progression as defined by IMWG criteria.
* Patients who are post auto-SCT as primary therapy must have received maintenance therapy with lenalidomide.
* Patients must be registered within 6 months of last dose of lenalidomide.
* Minimum of 3 months of maintenance therapy prior to disease progression.
* Age ≥ 18 years.
* Life expectancy of ≥12 weeks.
* KPS ≥ 70 or ECOG < 1 (Appendix IV)
* Patients must have adequate organ and marrow function as defined below:
* ANC ≥ 750/μL
* Platelets≥ 50,000/μL
* Total bilirubin ≤ 1.5 mg/dL
* AST(SGOT) ≤ 3 X upper limit of normal.
* ALT(SGPT) ≤ 3 X upper limit of normal.
* Cardiac Ejection Fraction ≥ 40%
* Serum Creatinine ≤ 2.0 mg/dL
* Patients must have an adequate number of CD34+ stem cells collected to allow for transplantation (defined as ≥ 2x10^6 CD34+ cells / kg body weight). If not previously collected and stored or if previous collection was inadequate, the patient must be willing to undergo stem cell mobilization and collection as per standard practice.
* Patients who participate in this study must be willing and able to tolerate prophylactic anticoagulation either with aspirin, low-molecular weight heparin (LMWH), or warfarin.
* Ability to understand and the willingness to sign a written informed consent document.
* Patient must be determined fit to undergo auto-SCT procedure by a study physician.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the POMALYST REMS™ program. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing pomalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.

  * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e.,has had menses at any time in the preceding 24 consecutive months).
* All study participants must be registered into the mandatory POMALYST REMS™ program, and be willing and able to comply with the requirements of the POMALYST REMS™ program.

  * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

* Patients who have had myeloma therapy within 14 days prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier. Patients may have received bisphosphonate therapy or radiation therapy as part of routine myeloma care at any time prior to study entry.
* Patients may not be receiving any other investigational agents.
* Any prior use of thalidomide or pomalidomide.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lenalidomide (including thalidomide) clarithromycin, or melphalan.
* Known prior positivity for active HIV or infectious hepatitis, type B or C.
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure , unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and lactating women are excluded from the study because the risks to an unborn fetus or potential risks in nursing infants are unknown.
* History of thrombosis or thromboembolic event within last 30 days prior to study entry.
* Patients with CNS involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-12; Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
overall response rate | at 9 months after the start of treatment
  Very Good PR or greater will be evaluated nine months postrandomization according to International Uniform Response Criteria.

SECONDARY OUTCOMES:
safety analyses | 3 years
  The frequency of subjects experiencing a specific adverse event will be tabulated overall and by each treatment course. In the by-subject analysis, a subject having the same event more than once will be counted only once. Adverse events will be summarized by worst NCI CTCAE grade. Laboratory data will be graded according to NCI CTCAE severity grade
overall survival | 1 year
progression free survival | 1 year
Determine the rates of ≥ Grade 3 toxicities | 1 year
  according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 as specified in section 10.0.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Giralt, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - North Shore LIJ, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - SUNY Upstate Medical University, Syracuse, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/